CLINICAL TRIAL: NCT02853539
Title: Denosumab Counteracts Metabolic Bone Disease in Chronic Intestinal Failure Patients: A Randomized, Controlled Clinical Trial
Brief Title: Denosumab in Metabolic Bone Disease in Chronic Intestinal Failure Patients
Acronym: Denoz
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Head of the Department, Stanley Dudrick's Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Denozumab
Record Dates: First submitted 2016-07-19; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Metabolic Bone Disease
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab (Experimental): One per 6 months subcutaneous injection of Denosumab (2 doses in total)
  Interventions: Drug: Denosumab
- No Denosumab (No Intervention): No intervention, just observation of HPN patients

INTERVENTIONS:
Drug: Denosumab — Subcutaneous injection of Denosumab
  Other Names: Prolia
  Arms: Denosumab

SUMMARY:
Low bone mineral density (BMD) is commonly reported in patients receiving home parenteral nutrition (HPN). Denosumab represent a new drug, which helped to prevent osteoclast. The aim of the study was to assess its value in chronic intestinal failure patients.

DETAILED DESCRIPTION:
Low bone mineral density (BMD) is commonly reported in patients receiving home parenteral nutrition (HPN). Oral and intravenous calcium, vitamin D and bisphosphonates have been commonly used to treat BMD, but their efficiency is may be inadequate due to limited absorption and compliance. Denosumab represent a new drug, which helped to prevent osteoclast development and activation, hence decreased bone resorption in some studies. The aim of the study was to assess its value in chronic intestinal failure patients receiving HPN.

Between November 2011 and March 2013 denosumab was administered to 16 HPN patients (9 F, 7 M mean age 55.4) with intestinal failure. Regional dual-energy x-ray absorptiometry of spine and hip were performed before the therapy was initiated, and after 12 months. BMD, T-score and Z-score were measured.

ELIGIBILITY:
Inclusion Criteria:

* intestinal failure requiring home parental nutrition
* bone disease measurement

Exclusion Criteria:

* intestinal failure not requiring HPN
* diagnostic modalities impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Improvement of bone structure: Spine | 36 months
  The increase of spine bone density measured by the change of Standard Deviation (SD) measured by DEXA at the level L1-L4
Improvement of bone structure: Femur | 36 months
  The increase of femur bone density measured by the change of Standard Deviation (SD) measured by DEXA at femur trochanter and shaft

SECONDARY OUTCOMES:
Treatment tolerance: gastrointestinal | 36 months
  The presence of adverse events from gastrointestinal tract: nausea, vomiting, diarhhoea
Treatment tolerance: bone pain | 36 months
  The presence of bone pain assessed with VAS score

CONTACTS AND LOCATIONS:
Locations (1):
- Stanley Dudrick's Memorial Hospital, Skawina, Poland

IPD SHARING:
Plan to Share IPD: Undecided